CLINICAL TRIAL: NCT03829930
Title: A Phase I Study of Entinostat in Combination With Enzalutamide for Treatment of Patients With Castration-Resistant Prostate Cancer
Brief Title: Combination of Entinostat and Enzalutamide in Advanced Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor discontinued the drug
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Jianqing Lin, Medical Oncologist, George Washington University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GWCC 1000
Record Dates: First submitted 2019-01-26; First posted 2019-02-04 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Prostate Adenocarcinoma
Keywords: Castration resistant prostate cancer
MeSH Terms: interventions — entinostat; enzalutamide

STUDY DESIGN:
Intervention Model Description: 3+3 Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entinostat and Enzalutamide (Experimental): Entinostat and Enzalutamide
  Interventions: Drug: Entinostat; Drug: Enzalutamide

INTERVENTIONS:
Drug: Entinostat — Entinostat is formulated for oral administration. A food effect is evident for entinostat; exposure is significantly reduced when entinostat is administered with a high fat meal. Accordingly, entinostat is to be administered on an empty stomach, at least 1 hour before and 2 hours after a meal. Entinostat tablets should not be split, crushed, or chewed. Consult the individual clinical protocols for specific dosing instructions.
  Dose level 1: 3mg PO weekly. Dose level 2: 5mg PO weekly.
  Other Names: SYND-275 amd MS-275
Drug: Enzalutamide — Dose level 1: 160 mg PO daily. Dose level 2: 160 mg PO daily.
  Other Names: MDV3100

SUMMARY:
To determine the safety and tolerability of Entinostat in combination with Enzalutamide in metastatic castrate resistant prostate cancer

DETAILED DESCRIPTION:
This study is designed to determine the safety and tolerability of Entinostat with Enzalutamide for treatment of patients with castration-resistant prostate cancer. There will be two dose levels of Entinostat in combination with same dose of Enzalutamide. Patients will be followed during treatment and 1 month post discontinuation.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Age >/= 18 years and are capable of giving informed consent. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patients must have a pathologically confirmed diagnosis of prostate adenocarcinoma. Features of neuroendocrine phenotype are allowed.
* Patients must have evidence of castration resistant metastatic disease and eligible for Enzalutamide per standard guidelines. Castration resistant non-metastatic disease is allowed in phase I study if subject is candidate for Enzalutamide.
* Patients must have and ECOG performance status of ≤ 2.(appendix D)
* Patients must be on continuous LHRH agonist or antagonist treatment or surgically castrated with castrate levels of testosterone (< 20 ng/dl).
* Any number of prior chemotherapy regimens are allowed. Chemotherapy naïve patients are allowed.
* If patient is already on Enzalutamide at a dose of 160mg daily, he is allowed if he can have baseline image and PSA within 1 month of the start of entinostat.
* Patients may have had androgen synthesis inhibitors or other investigational drugs. Patient must have discontinued flutamide or nilutamide or other AR targeted agents (including abiraterone) for at least 4 weeks and bicalutamide for at least 6 weeks prior to day 1 of treatment.
* Patients receiving treatment with bisphosphonates or denosumab must remain on treatment during the study.
* Patients must not require concurrent radiation or other chemotherapy while receiving protocol therapy. Patients may have received previous radiation but must have completed radiation at least 4 weeks (8 weeks for radiation to the brain) prior to registration.
* Patients must have recovered to grade ≤ 1 from all acute toxicity of previous radiation, hormonal or chemotherapy treatments.
* Patient agrees to use an acceptable method for contraception during the entire study treatment period through 4 months after the last dose of entinostat.
* Adequate renal function as defined by serum creatinine ≤ 1.5 x ULN. If creatinine >1.5 x ULN, calculated or measured creatinine clearance must be ≥ 60 mL/minute (Cockcroft-Gault).
* ANC > 1500/mm³, platelets > 100,000/mm³, Hgb > 9 g/dL.
* Total bilirubin ≤ ULN, SGOT (AST) and SGPT (ALT)< 1.5 x ULN. AST and/or ALT may be up to 5X ULN in the setting of known liver metastasis.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Patient was treated and discontinued Enzalutamide previously for any reason.
* Major surgery within 28 days or serious infection requiring IV antibiotics within 14 days preceding the first dose of study treatment
* Patient has received other investigational drugs within 14 days before enrollment.
* Known GI disease or GI procedure that could impact drug absorption in the upper bowel, or tolerance of Entinostat. Examples include but are not limited to partial gastrectomy, small bowel resection, pancreatectomy, malabsorption or celiac disease
* Ongoing nausea or vomiting of any severity without improvement after appropriate treatment.
* > Grade 1 diarrhea, not controlled with appropriate treatment.
* History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease requiring supplemental oxygen.
* Clinical and/or radiographic evidence of cerebral metastases. However, patients who have a history of central nervous system (CNS) metastasis but who have no radiographic or clinical evidence of residual tumor (eg, following complete surgical resection or stereotactic radiosurgery) are not excluded from participation in this study.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any EKG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Serious medical or psychiatric illness or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
* Any other currently active malignancy (excluding controlled non-melanoma skin cancer). Patients are considered NOT to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse.
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's Wort within 14 days prior to the first dose of Entinostat and during the study.
* History of seizure and on active therapy for seizure
* Known history of uncontrolled human immunodeficiency virus (HIV) infection. HIV positive patients will be allowed if they are on treatment and have an adequate CD4 count (CD4 count >200). Screening is not required in the absence of clinical findings or suspicion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Determination of a suitable dose of Entinostat in combination with Enzalutamide | 18 months
  Number of participants who experience an adverse event assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Progression Free Survival | 3 years
  Number of participants who survive without disease progression
Changes in circulating T cell subtype, peripheral blood mononuclear cell (PBMC) H3 acetylation, and phenotype of circulating Tregs | 18 months
  Analysis of immunomodulatory effects of Entinostat

CONTACTS AND LOCATIONS:
Overall Officials: Jianquig Lin, MD, Principal Investigator — George Washington Cancer Center
Locations (1):
- George Washington University - Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Lytton B. Prostate cancer: a brief history and the discovery of hormonal ablation treatment. J Urol. 2001 Jun;165(6 Pt 1):1859-62. No abstract available. PMID 11371867
- [Background] Carroll PR, Kantoff PW, Balk SP, Brown MA, D'amico AV, George DJ, Grossfeld GD, Johnson CS, Kelly WK, Klotz L, Lee WR, Lubeck DP, Mcleod DG, Oh WK, Pollack A, Sartor O, Smith MR, Hart C; Second International Conference on Newer Approaches to Androgen Deprivation Therapy (ADT) in Prostate Cancer. Overview consensus statement. Newer approaches to androgen deprivation therapy in prostate cancer. Urology. 2002 Sep;60(3 Suppl 1):1-6. doi: 10.1016/s0090-4295(02)01559-5. No abstract available. PMID 12231036
- [Background] Denis L, Murphy GP. Overview of phase III trials on combined androgen treatment in patients with metastatic prostate cancer. Cancer. 1993 Dec 15;72(12 Suppl):3888-95. doi: 10.1002/1097-0142(19931215)72:12+3.0.co;2-b. No abstract available. PMID 8252511
- [Background] Hellerstedt BA, Pienta KJ. The current state of hormonal therapy for prostate cancer. CA Cancer J Clin. 2002 May-Jun;52(3):154-79. doi: 10.3322/canjclin.52.3.154. PMID 12018929
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Small EJ, Schellhammer PF, Higano CS, Redfern CH, Nemunaitis JJ, Valone FH, Verjee SS, Jones LA, Hershberg RM. Placebo-controlled phase III trial of immunologic therapy with sipuleucel-T (APC8015) in patients with metastatic, asymptomatic hormone refractory prostate cancer. J Clin Oncol. 2006 Jul 1;24(19):3089-94. doi: 10.1200/JCO.2005.04.5252. PMID 16809734
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Knudsen KE, Scher HI. Starving the addiction: new opportunities for durable suppression of AR signaling in prostate cancer. Clin Cancer Res. 2009 Aug 1;15(15):4792-8. doi: 10.1158/1078-0432.CCR-08-2660. Epub 2009 Jul 28. PMID 19638458
- [Background] Nelson PS. Molecular states underlying androgen receptor activation: a framework for therapeutics targeting androgen signaling in prostate cancer. J Clin Oncol. 2012 Feb 20;30(6):644-6. doi: 10.1200/JCO.2011.39.1300. Epub 2011 Dec 19. No abstract available. PMID 22184375
- [Background] Tran C, Ouk S, Clegg NJ, Chen Y, Watson PA, Arora V, Wongvipat J, Smith-Jones PM, Yoo D, Kwon A, Wasielewska T, Welsbie D, Chen CD, Higano CS, Beer TM, Hung DT, Scher HI, Jung ME, Sawyers CL. Development of a second-generation antiandrogen for treatment of advanced prostate cancer. Science. 2009 May 8;324(5928):787-90. doi: 10.1126/science.1168175. Epub 2009 Apr 9. PMID 19359544
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] Beer TM, Tombal B. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Oct 30;371(18):1755-6. doi: 10.1056/NEJMc1410239. No abstract available. PMID 25354111
- [Background] Antonarakis ES, Lu C, Wang H, Luber B, Nakazawa M, Roeser JC, Chen Y, Mohammad TA, Chen Y, Fedor HL, Lotan TL, Zheng Q, De Marzo AM, Isaacs JT, Isaacs WB, Nadal R, Paller CJ, Denmeade SR, Carducci MA, Eisenberger MA, Luo J. AR-V7 and resistance to enzalutamide and abiraterone in prostate cancer. N Engl J Med. 2014 Sep 11;371(11):1028-38. doi: 10.1056/NEJMoa1315815. Epub 2014 Sep 3. PMID 25184630
- [Background] Lin J, Wang C, Kelly WK. Targeting epigenetics for the treatment of prostate cancer: recent progress and future directions. Semin Oncol. 2013 Jun;40(3):393-401. doi: 10.1053/j.seminoncol.2013.04.010. PMID 23806502
- [Background] Kaushik D, Vashistha V, Isharwal S, Sediqe SA, Lin MF. Histone deacetylase inhibitors in castration-resistant prostate cancer: molecular mechanism of action and recent clinical trials. Ther Adv Urol. 2015 Dec;7(6):388-95. doi: 10.1177/1756287215597637. PMID 26622323
- [Background] Gameiro SR, Malamas AS, Tsang KY, Ferrone S, Hodge JW. Inhibitors of histone deacetylase 1 reverse the immune evasion phenotype to enhance T-cell mediated lysis of prostate and breast carcinoma cells. Oncotarget. 2016 Feb 16;7(7):7390-402. doi: 10.18632/oncotarget.7180. PMID 26862729
- [Background] Gilbert J, Baker SD, Bowling MK, Grochow L, Figg WD, Zabelina Y, Donehower RC, Carducci MA. A phase I dose escalation and bioavailability study of oral sodium phenylbutyrate in patients with refractory solid tumor malignancies. Clin Cancer Res. 2001 Aug;7(8):2292-300. PMID 11489804
- [Background] Rathkopf D, Wong BY, Ross RW, Anand A, Tanaka E, Woo MM, Hu J, Dzik-Jurasz A, Yang W, Scher HI. A phase I study of oral panobinostat alone and in combination with docetaxel in patients with castration-resistant prostate cancer. Cancer Chemother Pharmacol. 2010 May;66(1):181-9. doi: 10.1007/s00280-010-1289-x. Epub 2010 Mar 9. PMID 20217089
- [Background] Saito A, Yamashita T, Mariko Y, Nosaka Y, Tsuchiya K, Ando T, Suzuki T, Tsuruo T, Nakanishi O. A synthetic inhibitor of histone deacetylase, MS-27-275, with marked in vivo antitumor activity against human tumors. Proc Natl Acad Sci U S A. 1999 Apr 13;96(8):4592-7. doi: 10.1073/pnas.96.8.4592. PMID 10200307
- [Background] Witta SE, Jotte RM, Konduri K, Neubauer MA, Spira AI, Ruxer RL, Varella-Garcia M, Bunn PA Jr, Hirsch FR. Randomized phase II trial of erlotinib with and without entinostat in patients with advanced non-small-cell lung cancer who progressed on prior chemotherapy. J Clin Oncol. 2012 Jun 20;30(18):2248-55. doi: 10.1200/JCO.2011.38.9411. Epub 2012 Apr 16. PMID 22508830
- [Background] Gore SD, Jiemjit A, Silverman LB, et al. Combined methyltransferase/histone deacetylase inhibition with 5-azacitidine and MS-275 in patients with MDS, CMMoL and AML: Clinical response, histone acetylation and DNA damage. Blood 2006; 108: Abstract 517
- [Background] Yardley DA, Ismail-Khan RR, Melichar B, Lichinitser M, Munster PN, Klein PM, Cruickshank S, Miller KD, Lee MJ, Trepel JB. Randomized phase II, double-blind, placebo-controlled study of exemestane with or without entinostat in postmenopausal women with locally recurrent or metastatic estrogen receptor-positive breast cancer progressing on treatment with a nonsteroidal aromatase inhibitor. J Clin Oncol. 2013 Jun 10;31(17):2128-35. doi: 10.1200/JCO.2012.43.7251. Epub 2013 May 6. PMID 23650416
- [Background] Shen L, Ciesielski M, Ramakrishnan S, Miles KM, Ellis L, Sotomayor P, Shrikant P, Fenstermaker R, Pili R. Class I histone deacetylase inhibitor entinostat suppresses regulatory T cells and enhances immunotherapies in renal and prostate cancer models. PLoS One. 2012;7(1):e30815. doi: 10.1371/journal.pone.0030815. Epub 2012 Jan 27. PMID 22303460
- [Background] Kato Y, Yoshino I, Egusa C, Maeda T, Pili R, Tsuboi R. Combination of HDAC inhibitor MS-275 and IL-2 increased anti-tumor effect in a melanoma model via activated cytotoxic T cells. J Dermatol Sci. 2014 Aug;75(2):140-7. doi: 10.1016/j.jdermsci.2014.04.014. Epub 2014 May 14. PMID 24866536
- [Background] Pili R, Salumbides B, Zhao M, Altiok S, Qian D, Zwiebel J, Carducci MA, Rudek MA. Phase I study of the histone deacetylase inhibitor entinostat in combination with 13-cis retinoic acid in patients with solid tumours. Br J Cancer. 2012 Jan 3;106(1):77-84. doi: 10.1038/bjc.2011.527. Epub 2011 Dec 1. PMID 22134508
- See also: NCT00859472 — https://clinicaltrials.gov/
- See also: NCT00878436 — https://clinicaltrials.gov/